CLINICAL TRIAL: NCT01324310
Title: A Phase I Open-label, 2-period Study to Evaluate the Influence of Multiple Oral Doses of Ketoconazole on the Single Dose Pharmacokinetics of Romidepsin in Subjects With Advanced Cancer
Brief Title: Influence of Ketoconazole on the Pharmacokinetics of Romidepsin in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ROMI-ADVM-001; 2010-022144-20 (EudraCT Number)
Record Dates: First submitted 2011-03-25; First posted 2011-03-29 (Estimated); Results first posted 2013-05-15 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Hematologic Malignancy; Malignant Lymphoma
Keywords: ROMI-001; romi; Romidepsin; Istodax; advanced malignancy; PK; pharmacokinetics
MeSH Terms: conditions — Hematologic Neoplasms; Lymphoma | interventions — romidepsin; Ketoconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Romidepsin and ketoconazole (Experimental): Romidepsin 8 mg/m^2 intravenous infused over 4 hours on Day 1 and Day 8.
  Ketoconazole 400 mg oral once daily on Days 4-8
  Interventions: Drug: Romidepsin; Drug: Ketoconazole

INTERVENTIONS:
Drug: Romidepsin — Romidepsin 8 mg/m^2 intravenous infused over 4 hours on Day 1 and Day 8.
  Other Names: Istodax®, Romi, ROMI
Drug: Ketoconazole — Ketoconazole 400 mg oral once daily on Days 4-8

SUMMARY:
The purpose of this study is to evaluate the effect and safety of multiple doses of ketoconazole on the pharmacokinetics of romidepsin after a single intravenous (IV) infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 18 years of age or older at the time of signing the informed consent document.
2. Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures are conducted.
3. Able to adhere to the study visit schedule and other protocol requirements.
4. Must have diagnosis of advanced malignancy and must have failed other available therapies considered standard of care for their disease.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
6. Negative urine or serum pregnancy test on females of childbearing potential; and
7. All females of childbearing potential must use an effective barrier method of contraception (either an intrauterine contraceptive device [IUCD] or double barrier method using condoms or a diaphragm plus spermicide) during the treatment period and for at least 1 month thereafter. Male subjects should use a barrier method of contraception during the treatment period and for at least 3 months thereafter. Female subjects should avoid the use of estrogen-containing contraceptives, since romidepsin may reduce the effectiveness of estrogen-containing contraceptives. An in vitro binding assay determined that romidepsin competes with β-estradiol for binding to estrogen receptors.

Exclusion Criteria:

1. Any significant medical condition or psychiatric illness that would prevent the subject from participating in the study.
2. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.
3. Subjects with significant gastrointestinal disease that may impair drug absorption, such as subjects with a history of Cohn's disease, colectomy, gastrectomy, celiac disease, or other diseases with known malabsorption.
4. Serum potassium < 3.8 mmol/L or serum magnesium < 0.85 mmol/L (magnesium converts to 2.1 mg/dl or 1.7 mEq/L) (electrolyte abnormalities can be corrected with supplementation to meet inclusion criteria).
5. Concomitant use of drugs that may cause a significant prolongation of the corrected measurement of the time between the start of the cardiac Q wave and the end of the T wave (QTc).
6. Concomitant use of Cytochrome P 450 3A4 (CYP3A4) strong inhibitors within 1 week of trial medications.
7. Concomitant use of CYP3A4 strong inducers within 2 weeks of trial medications.
8. Concomitant use of therapeutic warfarin due to a potential drug interaction. Use of a low dose of warfarin or another anticoagulant to maintain patency of venous access port and cannulas is permitted.
9. Clinically significant active infection.
10. Known infection with Human Immunodeficiency Virus (HIV), hepatitis B, or hepatitis C.
11. Inadequate bone marrow or other organ function as evidenced by:

    * Hemoglobin < 9 g/dL (transfusions and/or erythropoietin are permitted);
    * Absolute neutrophil count (ANC) ≤ 1.0 * 10^9 cells/L [subjects with neutropenia (ANC 1-1.5) as a function of their disease may be supported with granulocyte-colony stimulating factor (G-CSF)];
    * Platelet count < 100 * 10^9 cells/L or platelet count < 75 * 10^9 cells/L if bone marrow disease involvement is documented;
    * Total bilirubin > 1.5 * upper limit of normal (ULN) or > 2.0 * ULN in the presence of demonstrable liver metastases;
    * Serum aspartate transaminase/serum glutamic oxaloacetic transaminase (AST/SGOT) and alanine transaminase/serum glutamic pyruvic transaminase (ALT/SGPT) > 1.5 * ULN or > 2.0 * ULN in the presence of demonstrable liver metastases; or
    * Serum creatinine > 2.0 * ULN;
12. Prior chemotherapy treatment within 3 weeks prior to the first day of romidepsin treatment (6 weeks for nitrosoureas) or prior treatment with an investigational agent within 4 weeks prior to the first day of romidepsin treatment.
13. Prior radiotherapy within 4 weeks prior to the first day of treatment. Subjects who have not fully recovered or whose acute toxicity related to prior radiotherapy has not returned to baseline are ineligible.
14. Major surgery within 2 weeks of study entry (day 1).
15. Concomitant use of any other anti-cancer therapy.
16. Concomitant use of any investigational agent.
17. Prior exposure to romidepsin (other histone deacetylase[HDAC] inhibitors are allowed).
18. Any known cardiac abnormalities, such as:

    * Congenital long measure of the time between the start of the Q wave and the end of the T wave (QT) syndrome;
    * . Mean QTc formula (QTcF) interval > 450 msec;
    * A myocardial infarction within 12 months of study entry;
    * A history of coronary artery disease (CAD), e.g., angina Canadian Class II-IV. A stress imaging study should be performed for any subject whose cardiac status is uncertain. If abnormal, an angiography should be completed to define whether or not CAD is present.
    * An electrocardiogram (ECG) recorded at screening showing evidence of cardiac ischemia (ST depression of ≥ 2 mm, measured from isoelectric line to ST segment). A stress imaging study should be performed for any subject whose cardiac status is uncertain. If abnormal, an angiography should be completed to define whether or not CAD is present.
    * Congestive Heart Failure (CHF) that meets the New York Heart Association (NYHA) Class II to IV definitions (see Appendix F) and/or ejection fraction < 40% by multi gated acquisition (MUGA) scan or < 50% by echocardiogram and/or magnetic resonance imaging (MRI);
    * A known history of sustained ventricular tachycardia(VT), ventricular fibrillation (VF), torsades de pointes, or cardiac arrest unless currently addressed with an automatic implantable cardioverter defibrillator (AICD);
    * Hypertrophic cardiomegaly or restrictive cardiomyopathy from prior treatment or other causes (if in doubt, see ejection fraction criteria above);
    * Uncontrolled hypertension, i.e., blood pressure (BP) of ≥ 160/95; or
    * Any cardiac arrhythmia requiring anti-arrhythmic medication
19. Subjects who are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-04-01 (Actual); Primary Completion 2012-01-01 (Actual); Study Completion 2012-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ken Takeshita, MD, Study Director — Celgene Corporation
Locations (3):
- United States (2):
  - Florida Cancer Specialists, Sarasota, Florida
  - Sarah Cannon Research Institute, Nashville, Tennessee
- Sarah Cannon Research UK, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period occured over 6 months; the first participant enrolled on 01 July 2011; the last participant completed was 04 Jan 2012; 3 participating sites were involved (2 sites from the US and 1 in the UK); Overall, 15 subjects with advanced cancer were enrolled to ensure there was a minimum of 12 evaluable subjects
Groups:
- Romidepsin and Ketoconazole: Romidepsin 8 mg/m^2 intravenous infused over 4 hours on Day 1 and Day 8
  Ketoconazole 400 mg oral once daily on Days 4-8
Period: Overall Study
Arm/Group | Romidepsin and Ketoconazole
Started | 15
Completed | 13
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Disease Progression | 1

BASELINE CHARACTERISTICS:
Arm/Group | Romidepsin and Ketoconazole
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (11.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 12
  Asian | 2
  Black or African American | 0
  Other | 1
Region of Enrollment [Number; unit: Participants]
  United Kingdom | 6
  United States | 9
Height [Mean (Standard Deviation); unit: Centimeters] | 174.9 (9.59)
Weight [Mean (Standard Deviation); unit: kilograms] | 78.4 (18.77)
Body Surface Area (BSA) [Mean (Standard Deviation); unit: m^2] | 1.9 (0.24)
Eastern Cooperative Oncology Group Performance Status (ECOG) [Number; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status is used by doctors and researchers to assess how a patient's disease is progressing, assess how the disease affects the daily living activities of the patient and determine appropriate treatment and prognosis.
  0 = Fully Active (Most Favorable Activity); 1 = Restricted activity but ambulatory; 2 = Ambulatory but unable to carry out work activities; 3 = Limited Self-Care; 4 = Completely Disabled, No self-care
  Participants
    0 = Fully Active | 7
    1 = Restricted in physical strenuous activity | 8
    2 = Ambulatory but unable to work | 0
    3 = Limited Self Care | 0
    4 = Completely Disabled | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration Time-curve From Time 0 to the Time of the Last Quantifiable Concentration (AUC0-t)of Romidepsin
Description: AUC0-t: area under the plasma concentration time-curve from Time 0 to the time of the last quantifiable concentration (Ct), calculated by linear trapezoidal method when concentrations are increasing and the logarithmic trapezoidal method when concentrations are decreasing. For AUC0-t, an analysis of variance (ANOVA) model was used to estimate the ratio of geometric means and its 90% CI between romidepsin alone and romidepsin in the presence to ketoconazole.
Time Frame: Days 1 and 8; at 0 (pre-dose) 1, 2, 3, and 4 hours (end of infusion) and at 4.25, 4.5, 5, 6, 8, 10, 12, 24 and 48 hours after the initiation of IV infusion.
Population: Assessment on the influence of multiple doses of ketoconazole on the Pharmacokinetic (PK) of romidepsin; the PK population included participants who received at least 1 dose of study drug and had evaluable PK profiles. The reasons for study discontinuation: 1 subject withdrew due to an AE while another subject had disease progression.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- Romidepsin Day 1: Romidepsin 8 mg/m^2 intravenous infused over 4 hours on Day 1
- Romidepsin and Ketoconazole Day 8: Romidepsin 8 mg/m^2 intravenous infused over 4 hours on Day 8; Ketoconazole 400 mg oral once daily on Days 4-8
Arm/Group | Romidepsin Day 1 | Romidepsin and Ketoconazole Day 8
Number analyzed (Participants) | 15 | 13
ng*hr/mL | 911.0 (76.0) | 1020.7 (56.4)
Statistical Analysis 1: Comparison: Romidepsin Day 1 vs Romidepsin and Ketoconazole Day 8; Test type: Superiority or Other; ANOVA; Ratio of Geometric Mean = 124.4, 90% CI 2-sided [110.2 to 140.5] — Geometric means ratio ("Romidepsin + Ketoconazole"/"Romidepsin") and 90% CI of the ratio of geometric means are from an ANOVA model with treatment as fixed effect and subject as random effect on the natural log transformed PK values

2. Primary Outcome: Area Under the Plasma Concentration Time-curve From Time 0 to 24-hour (AUC 0-24)
Description: AUC 0-24: area under the plasma concentration time-curve from Time 0 to 24 hours, calculated by linear trapezoidal method when concentrations are increasing and the logarithmic trapezoidal method when concentrations are decreasing; for AUC 0-24 an analysis of variance (ANOVA) model was used to estimate the ratio of geometric means and its 90% confidence interval (CI) between romidepsin alone and romidepsin in the presence of ketoconazole
Time Frame: Days 1 and 8; at 0 (predose), 1, 2, 3, and 4 hours (end of infusion) and at 4.25, 4.5, 5, 6, 8, 10, 12, 24 and 48 hours after the initiation of IV infusion
Population: Assess the influence of multiple doses of ketoconazole on the pharmacokinetic (PK) of romidepsin; the PK population included participants who received at least 1 dose of study drug and had evaluable PK profiles. The reasons for study discontinuation: 1 subject withdrew due to an AE while another subject had disease progression.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Romidepsin Day 1 | Romidepsin and Ketoconazole Day 8
Number analyzed (Participants) | 15 | 13
ng*hr/mL | 900.1 (76.1) | 1002.2 (56.2)
Statistical Analysis 1: Comparison: Romidepsin Day 1 vs Romidepsin and Ketoconazole Day 8; Test type: Superiority or Other; ANOVA; Ratio of the Geometric Mean = 123.7, 90% CI 2-sided [109.6 to 139.6]

3. Primary Outcome: Area Under the Plasma Concentration Time-curve From Time 0 Extrapolated to Infinity (AUC0-∞)
Description: AUC0-∞: area under the plasma concentration time-curve from Time 0 extrapolated to infinity, calculated as [AUCt + Ct/λz].
Time Frame: Days 1 and 8; at 0 (pre-dose), 1, 2, 3, and 4 hours (end of infusion) and at 4.25, 4.5, 5, 6, 8, 10, 12, 24 and 48 hours after the initiation of IV infusion.
Population: Assess the influence of multiple doses of ketoconazole on the PK of romidepsin. The PK population included participants who received at least 1 dose of study drug and had evaluable PK profiles. The reasons for study discontinuation: 1 subject withdrew due to an AE while another subject had disease progression.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Romidepsin Day 1 | Romidepsin and Ketoconazole Day 8
Number analyzed (Participants) | 15 | 13
ng*hr/mL | 915.3 (75.9) | 1027.6 (59.3)
Statistical Analysis 1: Comparison: Romidepsin Day 1 vs Romidepsin and Ketoconazole Day 8; Test type: Superiority or Other; ANOVA; Ratio of the Geometric Mean = 124.6, 90% CI 2-sided [109.0 to 142.4]

4. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: Cmax: maximum observed plasma concentration, obtained directly from the observed concentration versus time data; for Cmax, an analysis of variance (ANOVA) model was used to estimate the ratio of geometric means and its 90% confidence interval (CI) between romidepsin alone and romidepsin in the presence of ketoconazole
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Romidepsin Day 1 | Romidepsin and Ketoconazole Day 8
Number analyzed (Participants) | 15 | 13
ng/mL | 229.05 (76.1) | 224.79 (45.2)
Statistical Analysis 1: Comparison: Romidepsin Day 1 vs Romidepsin and Ketoconazole Day 8; Test type: Superiority or Other; ANOVA; Ratio of the Geometric Mean = 109.5, 90% CI 2-sided [94.9 to 126.4]

5. Primary Outcome: Time to Maximum Observed Plasma Concentration (Tmax)
Description: Tmax: time to maximum observed Tmax, obtained directly from the observed concentration versus time data
Time Frame: as for outcome 3
Population: Assess the influence of multiple doses of ketoconazole on the PK of romidepsin; the PK population included participants who received at least 1 dose of study drug and had evaluable PK profiles. The reasons for study discontinuation: 1 subject withdrew due to an AE while another subject had disease progression.
Measure: Median (90% Confidence Interval); unit: hours
Arm/Group | Romidepsin Day 1 | Romidepsin and Ketoconazole Day 8
Number analyzed (Participants) | 15 | 13
hours | 3.257 (1.98,4.62) [1.98 to 4.62] | 2.992 (0.92,4.50) [0.93 to 4.50]
Statistical Analysis 1: Comparison: Romidepsin Day 1 vs Romidepsin and Ketoconazole Day 8; Note: The median, median difference ("romidepsin + ketoconazole" minus "romidepsin") and 90% CI of the median difference are from Hodges-Lehmann Estimate. The P-value is from Wilcoxon signed-rank test; Test type: Superiority or Other; p = 0.7422, Wilcoxon signed- rank; Median Difference (Final Values) = 0, 90% CI 2-sided [-0.485 to 0.095]

6. Primary Outcome: Estimate of the Terminal Elimination Half-life in Plasma (t1/2)
Description: Terminal elimination half-life (t1/2) in plasma, was calculated as [(ln 2)/λz]
Time Frame: Days 1 and 8; at 0 (pre-dose),1, 2, 3, and 4 hours (end of infusion) and at 4.25, 4.5, 5, 6, 8, 10, 12, 24 and 48 hours after the initiation of IV infusion.
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Romidepsin Day 1 | Romidepsin and Ketoconazole Day 8
Number analyzed (Participants) | 15 | 13
hours | 9.69 (26.4) | 10.171 (15.5)

7. Primary Outcome: Apparent Total Plasma Clearance (CL)
Description: Apparent total plasma clearance, (CL) calculated as [Dose/AUC 0-∞].
Time Frame: as for outcome 3
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Romidepsin Day 1 | Romidepsin and Ketoconazole Day 8
Number analyzed (Participants) | 15 | 13
L/hr | 16.922 (77.7) | 14.84 (63)

8. Primary Outcome: Apparent Total Volume of Distribution (Vz)
Description: Vz: apparent total volume of distribution, calculated as [(CL)/λz].
Time Frame: Days 1 and 8, At 0 (predose), 1, 2, 3, and 4 hours (end of infusion) and at 4.25, 4.5, 5, 6, 8, 10, 12, 24 and 48 hours after the initiation of IV infusion.
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Romidepsin Day 1 | Romidepsin and Ketoconazole Day 8
Number analyzed (Participants) | 15 | 13
Liter | 236.4 (88.7) | 217.78 (80.5)

9. Secondary Outcome: Summary of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: All 15 subjects in the safety population received at least 1 dose of romidepsin. AEs were considered related if assessed by the Investigator as possibly, probably or definitely related to study drug. Serious AEs (SAEs) are those that resulted in death, were life-threatening, required or prolonged inpatient hospitalization, resulted in persistent or significant disability/incapacity, congenital anomaly, or resulted in an important medical event that may have jeopardized the patient or required medical or surgical intervention to prevent one of the outcomes listed above.
Time Frame: Day 1 up to Day 36 (28 days after last treatment)
Population: The safety population consisted of all participants who received at least 1 dose of study drug. The Day 8 analysis population included 13 participants because two participants discontinued from the study prior to Day 8 (one due to an AE, the other due to disease progression).
Measure: Number; unit: participants
Groups:
- Romidepsin Plus Ketoconazole: Romidepsin 8 mg/m2 intravenous infused over 4 hours on Day 1 and Day 8. Ketoconazole 400 mg oral once daily on Days 4-8
Arm/Group | Romidepsin Plus Ketoconazole
Number analyzed (Participants) | 15
participants
  = > 1 TEAE | 15
  = > 1 TEAE related to any study drug | 14
  = > 1 TEAE related to Romidepsin | 14
  = > 1 TEAE related to Ketoconazole | 4
  = > 1 Serious TEAE | 4
  = > 1 Serious TEAE related to any drug | 1
  = > 1 Serious TEAE related to Romidepsin | 1
  = > 1 Serious TEAE related to Ketoconazole | 0
  = > 1 TEAE leading to discontinuation | 1
  = > 1 TEAE related discontinuation due to any drug | 0
  = > 1 Romidepsin related TEAE discontinuation | 0
  = > 1 Ketoconazole related TEAE discontinuation | 0
  Participants who died | 3

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 36 (28 days after last treatment)
Groups:
- Romidepsin Plus Ketoconazole: Romidepsin 8 mg/m^2 intravenous infused over 4 hours on Day 1 and Day 8. Ketoconazole 400 mg oral once daily on Days 4-8
Arm/Group | Romidepsin Plus Ketoconazole
Serious Adverse Events (participants affected / at risk) | 4/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Romidepsin Plus Ketoconazole (N=15)
General Physical Health Deterioration (General disorders) | 2
Pneumonia (Infections and infestations) | 2
Atrial Fibrillation (Cardiac disorders) | 1
Bile Duct Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Romidepsin Plus Ketoconazole (N=15)
Nausea (Gastrointestinal disorders) | 11
Vomiting (Gastrointestinal disorders) | 8
Constipation (Gastrointestinal disorders) | 3
Abdominal Pain Upper (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Intestinal Obstruction (Gastrointestinal disorders) | 1
Retching (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 7
Asthenia (General disorders) | 2
Chest Discomfort (General disorders) | 1
Chills (General disorders) | 1
Oedema Peripheral (General disorders) | 1
Pyrexia (General disorders) | 1
Decreased Appetite (Metabolism and nutrition disorders) | 8
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Headache (Nervous system disorders) | 5
Dysgeusia (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 1
Neuropathy Peripheral (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1
Confusional State (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Mental Status Changes (Psychiatric disorders) | 1
Urinary Tract Infection (Infections and infestations) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 1
Phlebitis (Vascular disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal Failure Acute (Renal and urinary disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There IS an agreement between the Principal Investigator and the Sponsor that restricts the PIs rights to publish trial results after the trial is completed. Upon investigator submission of a publication to Celgene, Celgene will complete its review within 60 days after receipt of the publication. Upon Celgene's request, the publication shall be delayed up to 90 additional days to enable Celgene to secure intellectual property protection that would be affected by such proposed publication.